CLINICAL TRIAL: NCT05514470
Title: Impact of Loss-of-function Mutations of Genes Encoding Cytosolic Aminoacyl-tRNA Synthetases on Protein Translation and Responses to Cellular Stress
Brief Title: Impact of Mutations in Aminoacyl tRNA Synthetases on Protein Translation and Cellular Stress
Acronym: FIBROMARS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study could not begin
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP220276; 2024-A01311-46 (Other: ID-RCB number)
Record Dates: First submitted 2022-06-17; First posted 2022-08-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Interstitial Lung and Liver Disease; Infantile Liver Failure Syndrome 1; Neurologic, Endocrine and Pancreatic Disease, Multisystem, Infantile-Onset 2; Rajab Interstitial Lung Disease With Brain Calcifications 2
Keywords: Cytosolic aminoacyl-tRNA synthetase; Mutations in the MARS1 gene; Mutations in the LARS1 gene; Mutations in the YARS1 gene; Mutations in the FARSA gene
MeSH Terms: conditions — Liver Diseases; Neurologic Manifestations; Pancreatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Patients with mutations in genes encoding cytosolic aminoacyl-tRNA synthetases and cared at Necker Hospital.
  Interventions: Other: Skin biopsy

INTERVENTIONS:
Other: Skin biopsy — A skin biopsy performed on the forearm or thigh depending on the patient's age and wishes, with a biopsy punch with a diameter of 3 to 4 mm depending on the child's age (3 for children under 3 years, 4 beyond).
  Culture of fibroblasts and immortalization.

SUMMARY:
Mutations in the genes encoding cytosolic aminoacyl-tRNA synthetases are responsible for early-onset multisystemic diseases including to varying degrees interstitial lung disease, liver damage, neurological and digestive disorders, and systemic inflammation. These are rare and severe diseases whose pathophysiology is poorly understood.

The investigative team hypothesizes that mutations within these genes are responsible for a decrease in protein translation and lead to a cellular stress response similar to that induced by amino acid deprivation. The investigative team also hypothesizes that these alterations could be corrected by high-dose supplementation in the culture medium of the corresponding amino acid.

The main objective of the study is to precisely determine the consequences of cytosolic aminoacyl-tRNA synthetase mutations at the cell level on protein translation.

DETAILED DESCRIPTION:
Mutations in the genes encoding cytosolic aminoacyl-tRNA synthetases are responsible for early-onset multisystemic diseases including to varying degrees interstitial lung disease, liver damage, neurological and digestive disorders, and systemic inflammation. These are rare and severe diseases whose pathophysiology is poorly understood.

The investigative team hypothesizes that mutations within these genes are responsible for a decrease in protein translation and lead to a cellular stress response similar to that induced by amino acid deprivation. The investigative team also hypothesizes that these alterations could be corrected by high-dose supplementation in the culture medium of the corresponding amino acid.

The main objective of the study is to precisely determine the consequences of cytosolic aminoacyl-tRNA synthetase mutations at the cell level on protein translation.

The parameters below will be studied in vitro in cell culture from skin biopsies of patients and control cells:

* Determination of total protein content
* The incorporation of d-methionine, leucine, tyrosine or phenylalanine into proteins
* The study of polysomes profiling
* The study of the assembly of the ribosomal 43S pre-initiation complex
* The phosphorylation of eIF2α and 4EBP and the expression of ATF4
* Ribosome profiling
* Transfer RNA (tRNA) sequencing
* The production of reactive oxygen species (ROS)

The results of these studies will be compared:

* Between patient cells and control cells
* Between genetically corrected patient cells, by stable transfection of the wild-type cDNA of the concerned genes and uncorrected cells
* Between patient cells cultured in medium enriched with the corresponding amino acid.

ELIGIBILITY:
Inclusion Criteria:

* Patients carrying mutations in genes encoding cytosolic aminoacyl-tRNA synthetases responsible for a multi-systemic phenotype
* Information and consent of the patient if an adult and of the holders of parental authority if a minor patient and of the minor patient

Exclusion Criteria:

- Non-consent of one of the holders of parental authority or of the minor patient or of adult patient

Contrôl patients :

* Fibroblasts from control patients without mutation in genes encoding cytosolic aminoacyl-tRNA synthetases, from an existing biological collection. The control patients will be selected according to the age at which the skin biopsy was performed in order to have an age match between the patients and the controls.
* Information and consent of the patient if an adult and of the holders of parental authority if a minor patient and of the minor patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Determination of total protein content | Day 0
  Determination of total protein content by Bicinchoninic acid assay.
Incorporation of d-methionine and d-phenylalanine into proteins | Day 0
  Incorporation of methionine and phenylalanine by labelled amino-acid fluorescent assays using ready-to-use kits.
Study of polysomes profiling | Day 0
  Study of polysome profils by differential sedimentation on sucrose gradients.
Study of the assembly of the ribosomal 43S pre-initiation complex | Day 0
  Study of the assembly of the ribosomal 43S pre-initiation complex by co-immunoprecipitation experiments.
Phosphorylation of eIF2α and 4EBP and the expression of ATF4 | Day 0
  Phosphorylation of eIF2α and 4EBP and the expression of ATF4 by western blot.
Ribosome profiling | Day 0
  Ribosome profiling by high throughput sequencing.
Transfer RNA (tRNA) sequencing | Day 0
  Transfer RNA (tRNA) sequencing by high throughput sequencing.
Production of reactive oxygen species (ROS) | Day 0
  Production of reactive oxygen species (ROS) by fluorescent measurement after cells' incubation with 2',7'- dichlorodihydrofluorescein diacetate (H2DCFDA).

CONTACTS AND LOCATIONS:
Overall Officials: Alice HADCHOUEL, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Isabelle SERMET-GAUDELUS, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No